CLINICAL TRIAL: NCT01383109
Title: A Human Mass Balance Study of Pyronaridine Using Accelerator Mass Spectrometry
Brief Title: Human Mass Balance Study of Pyronaridine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Shin Poong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-C-012-11
Record Dates: First submitted 2011-06-22; First posted 2011-06-28 (Estimated); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-11

CONDITIONS: Malaria
Keywords: Mass Balance; Accelerated Mass Spectrometry (AMS); microdose; Focus of the study: ADME
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pyronaridine (Experimental): All subjects will receive a single dose of Pyronaridine
  Interventions: Drug: 14C-labeled Pyronaridine

INTERVENTIONS:
Drug: 14C-labeled Pyronaridine — Single dose of 720 mg Pyronaridine together with 14C-Pyronaridine (approx. 100 µg, 800 nCi).

SUMMARY:
The combination of pyronaridine and artesunate is an antimalarial therapy in development. This mass balance study is intended to determine the rate and extent of excretion of total radioactivity in urine and feces following administration of a single oral micro-dose of 14C-pyronaridine in humans.

DETAILED DESCRIPTION:
This is a monocenter, open-label, non-placebo-controlled, single-group, single-dose study. Six male subjects will receive a single dose of Pyronaridine 720 mg orally administered together with 14C-Pyronaridine (approx. 100 µg, 800 nCi (29600 Bq)).

Safety measurements (12-lead ECG, vital signs, blood chemistry and haematology) and adverse events will be monitored throughout the study. Subjects will come to the clinic the evening before the dosing of Pyronaridine. After the drug intake at day 1, subjects will have regular in-house periods for specimen collection up to 87 days after the drug administration. Blood, feces and urine will be collected during the hospitalisation periods. Samples will be analyzed for radioactivity by Accelerator Mass Spectrometry (AMS).

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects between the ages of 40 and 55 years with a body weight between 60 and 90 kg and a body mass index calculated using Quetelet's Index - weight (kg)/height2 (m2) between 18.5 - 30.0
2. Signed and dated written informed consent form (ICF) before undergoing any study related activities, including discontinuation of any prohibited medications
3. Medically normal subjects with no significant abnormal findings at the screening physical examination as evaluated by the investigator
4. Strictly normal values of ALT, AST and bilirubin and normal or abnormal and clinically insignificant results (if agreed by the Investigator and the Sponsor on a case by case evaluation) of the other blood and urine laboratory parameters at screening
5. All sexually active male subjects and their partners are willing to undergo contraception as follows:

   All male subjects, including those who are sterilised (i.e., vasectomy), should use a condom. Their female partner must also use at least 1 of the medically acceptable forms of contraceptives listed below. Male subjects must not donate sperm or have unprotected sex during the study and until 87 days after taking the dose of investigational product.

   Medically acceptable contraceptives for this study are:

   Condoms in addition to:
   * Intrauterine devices
   * Hormonal contraceptives (oral, depot, patch, injectable, or vaginal ring)
   * Diaphragms with spermicidal cream or gel
   * Cervical cap with spermicidal cream or gel
   * Spermicidal foam
6. The ability to understand the requirements of the study and willingness to comply with all study procedures

Exclusion Criteria:

1. Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, acute QTc interval greater or equal to 450 mseconds), respiratory (including active tuberculosis), hepatic, renal, gastrointestinal, immunological (including active HIV-AIDS), neurological (including auditory), endocrine, infectious, malignancy, psychiatric or other clinical abnormality
2. Known history of hypersensitivity, allergic or adverse reactions to Pyronaridine
3. Known active Hepatitis A IgM (HAV-IgM), Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV Ab)
4. Seropositive HIV antibody
5. Previous participation in any clinical study with Pyramax
6. Presence or recent history (last two years) of tobacco abuse (≥10 cigarettes/day)
7. Known or suspected alcohol abuse or illicit drug use in the last 10 years before the study start or positive findings on urine drug screen
8. Intake of grapefruit and grapefruit juice alcoholic beverages or caffeine-containing food or beverages, such as coffee, tea, chocolate, or cola, 48 hours before study drug administration
9. Use of over-the-counter (OTC) medications, including vitamins, analgesics, or antacids, 1 week before the study start
10. Use of prescription medications 14 days before the study start or required chronic use of any prescription medication
11. Use of enzyme-altering agents (e.g., barbiturates, phenothiazines, cimetidine, etc.) within 30 days or 5 half lives, whichever the longer, before the study start
12. Plasma donation 1 month before the study start
13. Blood donation of 450 mL or more in the last 3 months before the study start
14. Participation in other clinical trials during the previous month in which an investigational drug or a commercially available drug was tested
15. Exposure to artificial ionizing radiation in the last 12 months (e.g., x-ray investigation, isotope studies)

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Borghini Fuhrer, PhD, Study Director — Medicines for Malaria Venture
Locations (1):
- Covance Clinical Research Unit AG, Allschwil, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pyronaridine
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all subjects who received a dose of the study drug.
Arm/Group | Pyronaridine
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6
Height [Mean (Standard Deviation); unit: cm] | 180.3 (8.2)
Weight [Mean (Standard Deviation); unit: kg] | 78.0 (7.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.1 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Analysis of 14C-Pyronaridine Total Radioactivity in Urine
Description: Radioactivity recovery in urine as a percent of the administered dose.
  Continuous collection of samples was performed through 168 hours post-dose, with intermittent 48 hour collections occurring thereafter
Time Frame: 2064 hours
Population: The pharmacokinetic population consisted of all subjects without any major violations of any inclusion or exclusion criteria, who received a dose of the study drug, had not received any unauthorised drug(s) which could have adversely affected the pharmacokinetic analysis, and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: % administered dose
Arm/Group | Pyronaridine
Number analyzed (Participants) | 6
% administered dose
  0-4h | 0.09 (0.02)
  4-8h | 0.16 (0.08)
  8-24h | 0.60 (0.20)
  24-48h | 0.71 (0.08)
  48-72h | 0.67 (0.24)
  72-96h | 0.63 (0.10)
  96-120h | 0.55 (0.08)
  120-144h | 0.55 (0.09)
  144-168h | 0.60 (0.23)
  168-336h | 3.87 (0.69)
  336-384h | 2.38 (0.60)
  384-504h | 2.38 (0.60)
  504-552h | 0.84 (0.37)
  552-672h | 1.81 (0.69)
  672-720h | 0.61 (0.23)
  720-840h | 1.34 (0.58)
  840-888h | 0.46 (0.23)
  888-1008h | 1.11 (0.45)
  1008-1056h | 0.42 (0.14)
  1056-1344h | 2.08 (0.61)
  1344-1392h | 0.27 (0.07)
  1392-1680h | 1.42 (0.34)
  1680-1728h | 0.20 (0.04)
  1728-2016h | 1.12 (0.26)
  2016-2064h | 0.17 (0.04)

2. Primary Outcome: Analysis of 14C-Pyronaridine Total Radioactivity in Feces
Description: Radioactivity recovery in feces as a percent of the administered dose.
  Continuous collection of samples was performed through 168 hours post-dose, with intermittent 48 hour collections occurring thereafter
Time Frame: 2064 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % administered dose
Arm/Group | Pyronaridine
Number analyzed (Participants) | 6
% administered dose
  24-48h | 7.31 (6.12)
  48-72h | 12.78 (8.45)
  72-96h | 5.83 (3.65)
  96-120h | 4.53 (1.68)
  120-144h | 2.11 (1.68)
  144-168h | 2.03 (2.13)
  168-336h | 7.89 (2.01)
  336-384h | 1.40 (0.78)
  384-504h | 2.69 (1.42)
  504-552h | 0.76 (0.39)
  552-672h | 1.58 (0.66)
  672-720h | 0.51 (0.17)
  720-840h | 1.01 (0.30)
  840-888h | 0.30 (0.11)
  888-1008h | 0.70 (0.31)
  1008-1056h | 0.26 (0.16)
  1056-1344h | 1.23 (0.53)
  1344-1392h | 0.15 (0.08)
  1392-1680h | 0.68 (0.13)
  1680-1728h | 0.09 (0.03)
  1728-2016h | 0.41 (0.18)
  2016-2064h | 0.07 (0.01)

3. Secondary Outcome: Total Radioactivity in Blood: AUC0-t, AUC0-∞
Description: Pharmacokinetic Parameters:
  AUC0-t: area under the plasma concentration-time curve from Hour 0 through the last quantifiable concentration time (LQCT), where LQCT is the time at which the last sample with a quantifiable concentration was collected AUC0-∞: area under the plasma concentration-time curve from Hour 0 to infinity
  PK sampling performed at predose, 0.5, 1, 2, 4, 8, 12 and 24 hours, and 2, 4, 6, 7, 14, 21, 28, 35 and 42 days post-dose
Time Frame: 42 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day*ng-eq/ml
Arm/Group | Pyronaridine
Number analyzed (Participants) | 6
day*ng-eq/ml
  AUC0-t | 1834 (530)
  AUC0-∞ | 3731 (1303)

4. Secondary Outcome: Total Radioactivity in Blood: Cmax
Description: Pharmacokinetic Parameters:
  Cmax: maximum observed peak observed concentration
  PK sampling performed at predose, 0.5, 1, 2, 4, 8, 12 and 24 hours, and 2, 4, 6, 7, 14, 21, 28, 35 and 42 days post-dose
Time Frame: 42 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-eq/ml
Arm/Group | Pyronaridine
Number analyzed (Participants) | 6
ng-eq/ml | 271 (113)

5. Secondary Outcome: Total Radioactivity in Blood: Half-life, Tmax
Description: Pharmacokinetic Parameters:
  Half-life: computed as ln (2) / Kel Tmax: time to maximum concentration
  PK sampling performed at predose, 0.5, 1, 2, 4, 8, 12 and 24 hours, and 2, 4, 6, 7, 14, 21, 28, 35 and 42 days post-dose
Time Frame: 42 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pyronaridine
Number analyzed (Participants) | 6
days
  Half-life | 33.5 (11.4)
  Tmax | 0.111 (0.111)

ADVERSE EVENTS:
Time Frame: 87 days
Description: The condition of each subject was monitored throughout the study. In addition, any signs and symptoms were observed and elicited at least once a day by open questioning, such as "How have you been feeling since you were last asked?". Subjects were also encouraged to report spontaneously any adverse events during the study.
Arm/Group | Pyronaridine
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyronaridine (N=6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Elevated liver enzymes (Investigations) | 1 (1) — Alanine aminotransferase increased Aspartate aminotransferase increased Gamma glutamyl transferase increased
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No